CLINICAL TRIAL: NCT06348303
Title: A Prospective, Randomized, Single-blind, Pilot Study to Assess Drowsiness, Cognition, and Fall Risk Following Oral Metaxalone 640 mg (M640) Versus Metaxalone 800 mg in Healthy Subjects"
Brief Title: Study to Assess Drowsiness, Cognition, Fall Risk After Metaxalone 640 mg and Metaxalone 800 mg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Primus Pharmaceuticals (Industry)
Collaborators: ClinOhio Research Services, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PMMD-01
Record Dates: First submitted 2024-03-30; First posted 2024-04-04 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants
MeSH Terms: interventions — metaxalone; Tablets

STUDY DESIGN:
Intervention Model Description: Each participant will be enrolled to two (2), single dose, study treatment arms in a crossover design. The treatments will occur consecutively with seven (7) days separating days of dosing.
Who Masked: Participant
Masking Description: Single mask of participants. Participants will be prevented from knowing product dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active 640 mg (Active Comparator): Metaxalone (M640) 640 mg tablet, a single-dose at visit 2 of 4 visits.
  Interventions: Drug: Metaxalone m640 mg oral tablet
- Active 800 mg (Active Comparator): Metaxalone 800 mg tablet, a single-dose at Visit 3 of 4 visits.
  Interventions: Drug: Metaxalone 800 mg oral tablet

INTERVENTIONS:
Drug: Metaxalone m640 mg oral tablet — Metaxalone partially micronized 640 mg tablet
  Other Names: m640
  Arms: Active 640 mg
Drug: Metaxalone 800 mg oral tablet — Metaxalone non-micronized 800 mg oral tablet
  Other Names: Skelaxin
  Arms: Active 800 mg

SUMMARY:
Every participant will receive Metaxalone in two (2) stages, one week after the other. A single dose of each Metaxalone dose will be taken one (1) time after a high fat meal which must be eaten within 30 minutes. Every participant will be given written tests to measure drowsiness, reaction time and thinking process and will also be asked to take walking tests to assess fall risk. Participation in this study will last approximately 2-4 weeks.

DETAILED DESCRIPTION:
The Screening-Baseline Visit will include vital signs and urine testing, and a discussion of medications and current medical history. Participants will be given written tests to measure drowsiness, reaction time and thinking process and will also be asked to take walking tests to assess fall risk.

Visit 2 approximately one to two (1 to 2) week(s) later will be the first dosing day (Arm 1) after eating the high fat meal. The testing from Baseline will be repeated four (4) hours after the medication dose is taken.

Visit 3 approximately one (1) week later will be the second dosing day (Arm 2) after eating the high fat meal. The testing from Baseline will be repeated four (4) hours after the medication dose is taken.

The End of Study safety visit will take place one (1) week after Visit 3 by phone with a discussion of any side effects from the drug, recent medications, and any illness or injury experienced since the previous visit. Participants will be given end of study and discharge instructions.

ELIGIBILITY:
Inclusion Criteria:

* Weigh at least 120 pounds at Screening
* Medically healthy with no clinically significant medical co-morbidities impact endpoints

Exclusion Criteria:

* Current use of any medications known to affect sleep-wake cycle.
* Known sleep disorder.
* Current use of cimetidine.
* Current use of a monoamine oxidase Inhibitor (MAOI), selective serotonin reuptake inhibitor (SSRI), selective norepinephrine reuptake inhibitor (SNRI), 5- hydroxytryptamine (5-HT) agonist or any drug that has the potential to affect the serotonergic neurotransmitter system (e.g. mirtazapine, trazodone, tramadol).
* Positive urine test for amphetamines, barbiturates, cocaine, opiates, benzodiazepines, or cannabinoids.
* Participants taking skeletal muscle relaxants or sedative hypnotics.
* Participants with gastrointestinal disease affecting absorption.
* Participants with severe hepatic or renal impairment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Percentage of participants unable to maintain Tandem Stand Position for more than 10 seconds (position 3 of the 4-Stage Balance Test). | Baseline, Visit 2 dosing (Day 1), Visit 3 dosing (Day 8)
  Validated 4-Stage Balance Test after completion of an FDA standardized high-fat meal. Place one foot in front of the other, heel touching toes.
Change from baseline of gait during a stopwatch timed, stand, and walk activity from a seated position along a 30 foot path | Baseline, Visit 2 dosing (Day 1), Visit 3 dosing (Day 8)
  Timed Up and Go with Triaxial Accelerometry
Change from baseline of correct number of steps taken on a fixed 4 inch wide, 9 feet long path | Baseline, Visit 2 dosing (Day 1), Visit 3 dosing (Day 8)
  Tandem Walk Test

SECONDARY OUTCOMES:
Change from baseline of participants' subjective report of drowsiness on a 10-point scale | Baseline, Visit 2 dosing (Day 1), Visit 3 dosing (Day 8)
  Karolinska Sleepiness Scale where 1 = extremely alert and 10 = extremely sleepy, can't keep awake
Change from baseline of reaction to stimulus by computer generated visual prompts measured in milliseconds | Baseline, Visit 2 dosing (Day 1), Visit 3 dosing (Day 8)
  Reaction Time Test (RTT)
Change from baseline of participants' reasoning ability to recognize differences in six (6) computer generated shapes for 30 minutes | Baseline, Visit 2 dosing (Day 1), Visit 3 dosing (Day 8)
  Creyos Cognitive Test
The number of product related adverse events experienced by participants from Visit 2 through Visit 4 | Visit 2 dosing (Day 1, Visit 3 dosing (Day 8), Visit 4 End of Study (Day 15)
  Adverse and Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: J Lukban, DO, Study Director — Primus Pharmaceuticals, Inc.
Locations (1):
- ClinOhio Research Institute, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No